CLINICAL TRIAL: NCT04152499
Title: A Phase I-II, First-in-Human Study of SKB264 in Patients With Locally Advanced Unresectable /Metastatic Solid Tumors Who Are Refractory to Available Standard Therapies
Brief Title: Phase I-II, FIH, TROP2 ADC, Advanced Unresectable/Metastatic Solid Tumors, Refractory to Standard Therapies (KL264-01)
Acronym: MK-2870-001
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Klus Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KL264-01
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-06

CONDITIONS: Epithelial Ovarian Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Urothelial Carcinoma; Non-Small Cell Lung Cancer; Small-Cell Lung Cancer; Endometrial Carcinoma; Head and Neck Squamous Cell Carcinoma; Breast Cancer; Cervical Cancer
Keywords: TROP2, ADC
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (11):
- Phase I: Dose Escalation (Experimental): Five dose levels have been selected for evaluation in the Phase I part of the study: 2, 4, 6, 9, and 12 mg/kg of SKB264
  Interventions: Drug: SKB264
- Phase II: Triple Negative Breast Cancer (Experimental): Histologically documented or cytologically , incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Epithelial Ovarian Cancer (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Non-Small Cell Lung Cancer (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma (Experimental): Histologically or cytologically documented, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Extensive-stage Small Cell Lung Cancer (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: HR+/ HER2- Breast Cancer (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Head and Neck Squamous Cell Carcinoma (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Endometrial carcinoma (Experimental): Histologically documented or cytologically, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Urothelial carcinoma (Experimental): Histologically or cytologically documented, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264
- Phase II: Cervical Cancer (Experimental): Histologically or cytologically documented, incurable, locally advanced or metastatic cancer
  Interventions: Drug: SKB264

INTERVENTIONS:
Drug: SKB264 — SKB264 is an Antibody Drug Conjugate (ADC) targeting TROP2 expressing cancer cells.
  Other Names: MK-2870; Sacituzumab Tirumotecan (Sac-TMT)

SUMMARY:
A Phase I-II, First-in-Human Study of SKB264 (Sac-TMT; MK-2870) in Patients with Locally Advanced Unresectable/Metastatic Solid Tumors who are refractory to Available Standard Therapies. Patient must have historically documented, incurable, locally advanced or metastatic cancer that are refractory to standard therapies of one of the following types:

1. Triple negative breast cancer
2. Epithelial ovarian cancer
3. Non-small cell lung cancer
4. Gastric adenocarcinoma/Gastroesophageal junction adenocarcinoma
5. Small cell lung cancer
6. HR+/ HER2-breast cancer
7. Head and neck squamous cell carcinoma
8. Endometrial carcinoma
9. Urothelial carcinoma
10. Cervical cancer

DETAILED DESCRIPTION:
This is an open label, Phase I-II, first in human (FIH) study for SKB264 as monotherapy in patients who have locally advanced unresectable or metastatic solid tumor that is refractory to all standard therapies. TROP2 (trophoblast antigen 2) assessments will not be performed prior to enrollment but it will be assessed retrospectively. Confirmation of TROP2 (trophoblast antigen 2) expression by immunohistology or other means is not required, but the Sponsor will request fresh tumor biopsy or tissue specimens from archived materials for determination of TROP2 (trophoblast antigen 2) expression retrospectively. The patient must be, in the judgment of the investigator, an appropriate candidate for experimental therapy whose tumor is refractory to standard therapies. Patients will receive study drug as a single IV infusion at the prescribed dose level at each administration. Cycles will continue until disease progression or unacceptable toxicity. The study is divided into 2 parts (Phase I and Phase II).

ELIGIBILITY:
Diagnosis and Main Criteria for Inclusion:

Inclusion Criteria:

Patients must meet the following criteria for inclusion into the study:

Phase I:

1. Patients must be able to provide documented voluntary informed consent.
2. Male or female patient aged 18-75 years.
3. Histologically documented, incurable, locally advanced or metastatic epithelial origin malignant cancer, priority to include but not limited to the following tumor types:

   Breast cancer Ovarian epithelial cancer Non-small cell lung cancer Gastric adenocarcinoma Small cell lung cancer Urothelial carcinoma Note: Confirmation of TROP2 expression by immunohistology or other means is not required, but the Sponsor will request tissue specimens from fresh or archived materials for determination of TROP2 expression.
4. Measurable disease by CT/MRI during dose escalation.
5. Patients should have an unresectable locally advanced or metastatic solid tumor that is refractory to standard therapies, or have no standard therapies, or standard treatment is not applicable at this stage.
6. Granulocyte count ≥ 1.5×109/L, platelet count ≥ 100×109/L, and hemoglobin ≥ 9 g/dL.
7. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5×ULN.
8. Serum bilirubin ≤ 1.5 mg/dL (Patients with known Gilbert disease who have serum bilirubin level ≤ 3 ×ULN may be enrolled)., aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 × upper limit of normal (ULN), with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) and patients with hepatic and/or bone metastases (alkaline phosphatase ≤ 5 × ULN).
9. Creatinine clearance ≥ 50 mL/min calculated by Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration, or Modification of Diet in Renal Disease formulas. Note that 24 hour urine collection is not required but is allowed.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
11. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception during study treatment. Female and male patient treated with SKB264 should continue contraception use for 7 months after the last dose. Such methods include combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.

    * Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug. The same rules are valid for male patients involved in this clinical trial if they have a partner of childbirth potential. Male patients must always use a condom.
    * Women are excluded from birth control if they had had tubal ligation or a hysterectomy.
12. Patients must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and vitiligo.
13. Expected survival ≥ 3 months.

Phase II:

1. Patients must be able to provide documented voluntary informed consent.
2. Male or female patient aged ≥ 18 years.
3. Histologically or cytologically documented, incurable, locally advanced, recurrent or metastatic cancer, including the following tumor types:

   * Cohort 1: triple negative breast cancer (< 1% expression for estrogen receptor [ER] and progesterone receptor [PR] and HER2 negative)
   * Cohort 2: ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
   * Cohort 3: non-small cell lung cancer
   * Cohort 4: gastric adenocarcinoma or gastroesophageal junction adenocarcinoma (HER2 negative)
   * Cohort 6: HR+/ HER2- breast cancer (≥1% expression for ER and/or PR and HER2 negative)
   * Cohort 7: Head and neck squamous cell carcinoma (including primary tumor location of oropharynx, oral cavity, hypopharynx, or larynx. Other primary tumor sites of HNSCC are not eligible)
   * Cohort 8: Endometrial carcinoma (including carcinosarcoma, but excluding sarcoma and neuroendocrine endometrial carcinoma)
   * Cohort 9: Urothelial carcinoma (including urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra, patients with mixed histology are eligible provided urothelial component > 50% and plasmacytoid component<10%, patients whose tumors contain any neuroendocrine component are not eligible)
   * Cohort 10: Cervical cancer (including squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix) Note: Evaluation of TROP-2 expression is required.
4. Measurable disease by CT/MRI.
5. Patients should have an unresectable locally advanced or metastatic solid tumor that is refractory to standard therapies.
6. Neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109/L, and hemoglobin ≥ 9 g/dL.
7. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5×ULN.
8. Serum bilirubin ≤ 1.5 ×ULN (Patients with known Gilbert disease who have serum bilirubin level ≤ 3 ×ULN may be enrolled), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 × upper limit of normal (ULN), with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) and patients with hepatic and/or bone metastases (alkaline phosphatase ≤ 5 × ULN).
9. Creatinine clearance ≥ 30 mL/min calculated by Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), or Modification of Diet in Renal Disease (MDRD) formulas. Note that 24 hour urine collection is not required but is allowed.
10. ECOG Performance Status 0 or 1.
11. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception during study treatment. Female and male patient treated with SKB264 should continue contraception use for 6 months after the last dose. Such methods include combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.

    * Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug. The same rules are valid for male patients involved in this clinical trial if they have a partner of childbirth potential. Male patients must always use a condom.
    * Women are excluded from birth control if they had had tubal ligation or a hysterectomy.
12. Patients must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and vitiligo. Note: Subjects with endocrine AE of any grade are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
13. Expected survival ≥ 3 months.

Exclusion Criteria:

Patients that meet the following criteria will be excluded from entry into the study:

Phase I:

1. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure (New York Heart Association) III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
2. Symptomatic brain metastases or any radiation or surgery for brain metastases within 1 months of first infusion of study drug.
3. Subjects with second primary cancers (except for cured in situ non-melanoma skin cancer and in situ cervical cancer with no relapse in the last 3 years).
4. Require supplemental oxygen for daily activities.
5. Documented Grade ≥ 2 peripheral neuropathy.
6. History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, corneal disease that prevents/delays corneal healing, macular degeneration.
7. Subjects previously treated with TROP 2 targeted therapies.
8. Any standard cancer therapy (e.g. chemotherapy, hormonal therapy, radiotherapy, immunotherapy, biologic therapy treatment, or therapy with traditional Chinese medicines approved for anti-tumor treatment, etc.) within 4 weeks or five half-lives, whichever is shorter, of first infusion of study drug.
9. Any experimental therapy within 4 weeks or five half-lives, whichever is shorter, of first infusion of study drug.
10. Any major surgical procedure within 4 weeks of first infusion of study drug.
11. Diagnosed active liver disease, including viral or other hepatitis, current or history of alcoholism, or cirrhosis.
12. Have known prior positive test results or medical history for human immunodeficiency virus.
13. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or diabetes (HbA1c ≥ 9.0%).
14. Subjects who require use of strong inhibitors or inducers of CYP3A4 at least 14 days prior to and throughout Study. Use of strong inhibitors or inducers of CYP3A4 is not allowed in this study. List of representative examples of strong inhibitors or inducers of CYP3A4 is provided in Appendix III.
15. Pregnancy or lactation.
16. Left ventricular ejection fraction < 45% determined by echocardiogram or multiple gated acquisition scan.
17. Resting QTc > 480 msec at baseline.
18. Ascites requiring paracentesis ≥1 per week.
19. Symptomatic pleural effusion (< 90% oxygen saturation).
20. Subjects with non-infectious interstitial lung diseases (ILD) or medical history of pneumonia requiring steroid treatments; severe pulmonary dysfunction caused by lung diseases.
21. New diagnosed thromboembolic events that requires therapeutic intervention over the last 6 months (patients with stable control of lower limb deep venous thrombosis are allowed).
22. The investigator considers other situations that patients are not appropriate to participate in this trial.

Phase II:

1. Any patient who was treated in the Phase I part of this study.
2. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure (New York Heart Association) III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
3. Subjects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or other active CNS metastases.
4. Patients with active second primary cancers (except for cured in situ non-melanoma skin cancer and in situ cervical cancer with no relapse in the last 3 years, or other malignant cancers that have been cured and no evidence of recurrence).
5. Require supplemental oxygen for daily activities.
6. Documented Grade ≥ 2 peripheral neuropathy.
7. History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, corneal disease that prevents/delays corneal healing, macular degeneration.
8. Patients previously treated with TROP 2 targeted therapies at any time for early stage or metastatic disease.
9. Any standard cancer therapy (e.g. chemotherapy, hormonal therapy, radiotherapy, immunotherapy, biologic therapy treatment, or therapy with traditional Chinese medicines approved for anti-tumor treatment, etc.) within 4 weeks or 5 half-lives, whichever is shorter, of first infusion of study drug.
10. Any experimental therapy within 4 weeks or 5 half-lives, whichever is shorter, of first infusion of study drug.
11. Any major surgical procedure within 4 weeks of first infusion of study drug.
12. Diagnosed active liver disease, including viral or other hepatitis, current or history of alcoholism, or cirrhosis.
13. Have known prior positive test results or medical history for human immunodeficiency virus.
14. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or diabetes (HbA1c ≥ 9.0%).
15. Subjects who require use of strong inhibitors or inducers of CYP3A4 at least 14 days prior to and throughout Study. Use of strong inhibitors or inducers of CYP3A4 is not allowed in this Study. List of representative examples of strong inhibitors or inducers of CYP3A4 is provided in Appendix III.
16. Pregnancy or lactation.
17. Left ventricular ejection fraction < 45% determined by echocardiogram or multiple gated acquisition scan.
18. Resting QTcF > 480 msec at baseline.
19. Ascites requiring paracentesis >1 per week.
20. Symptomatic pleural effusion (< 90% oxygen saturation).
21. History of interstitial lung diseases (ILD) or non-infectious pneumonitis requiring steroid treatments; severe pulmonary dysfunction caused by lung diseases.
22. New diagnosed thromboembolic events that requires therapeutic intervention over the last 6 months (patients with stable control of lower limb deep venous thrombosis are allowed).
23. Known allergic to any components of SKB264, including excipients (including polysorbate-20); or history of severe hypersensitivity to another biologic therapy.
24. The investigator considers other situations that patients are not appropriate to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) and Recommended Doses for Expansion (RDEs) | Assess up to 12 months
  To determine the maximum tolerated dose (MTD) and/or recommended doses for expansion (RDEs). RDEs will not exceed MTD.
Phase II: Objective Response Rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  To evaluate the objective response rate (ORR) [Complete Response (CR) + Partial Response (PR)] of SKB264 when administered intravenously (IV) as monotherapy at the RDEs to patients with metastatic or locally advanced unresectable tumors.

SECONDARY OUTCOMES:
Phase I: Dose Limiting Toxicities (DLTs) | Day 28 days after first infusion of study drug
  To determine the dose limiting toxicities (DLTs) of SKB264 when administered IV twice (on Days 1 and 15) every 2 weeks in 4 weeks (28 days) cycles as monotherapy to patients with metastatic or locally advanced unresectable tumors.
Phase I: Overall safety and tolerability profile | from the date of informed consent until 30 days after last infusion of study drug or begin a new anti cancer therapy, whichever occurs first
  Percentage of patients with adverse events (AEs), serious adverse events (SAEs), AEs with Grade ≥ 3 per NCI CTCAE v5.0, adverse events of Special Interest (AESI) and AEs related to study drug.
Phase I: Preliminary efficacy based on ORR (Objective Response Rate) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months
  ORR (Objective Response Rate) as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, which will be complete response (CR) + partial response (PR)
Phase I: Preliminary efficacy based on DOR(Duration of Response) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months
  To evaluate preliminary efficacy in patients treated with SKB264 as monotherapy based on DOR(Duration of Response).
Phase I: Preliminary efficacy based on PFS(Progression-Free Survival) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months
  To evaluate preliminary efficacy in patients treated with SKB264 as monotherapy based on PFS(Progression-Free Survival).
Phase I: Preliminary efficacy based on OS(Overall Survival) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months
  To evaluate preliminary efficacy in patients treated with SKB264 as monotherapy based on OS(Overall Survival)
Phase I: Percentage of patients with ADA formation to SKB264. | From Cycle 1 to Cycle 6 and End of Treatment(EOT), approximately 12 months
  To assess the incidence of anti-drug antibody (ADA) formation to SKB264.
Phase I: PK parameters for SKB264-ADC, SKB264 TAB, and free KL610023 payload. | From Cycle 1 to Cycle 6 and End of Treatment(EOT), approximately 12 months
  To characterize the PK of SKB264-ADC, SKB264 TAB, and free KL610023 payload, such as Cmax
Phase II: Overall safety and tolerability profile | from the date of informed consent until 30 days after last infusion of study drug or begin a new anti cancer therapy, whichever occurs first
  Percentage of patients with adverse events (AEs), serious adverse events (SAEs), AEs with Grade ≥ 3 per NCI CTCAE v5.0, adverse events of Special Interest (AESI) and AEs related to study drug.
Phase II: Efficacy based on DOR (Duration of Response) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months.
  To evaluate efficacy in patients treated with SKB264 as monotherapy based on DOR(Duration of Response)
Phase II: Efficacy based on PFS (Progression-Free Survival) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months.
  To evaluate efficacy in patients treated with SKB264 as monotherapy based on PFS (Progression-Free Survival)
Phase II: Efficacy based on OS (Overall Survival) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, approximately 12 months.
  To evaluate efficacy in patients treated with SKB264 as monotherapy based on OS (Overall Survival)
Phase II: Percentage of patients with ADA formation to SKB264. | From Cycle 1 to Cycle 6 and End of Treatment(EOT), approximately 12 months
  To obtain Percentage of patients with ADA formation to SKB264.
Phase II: PK parameters for SKB264-ADC, SKB264 TAB, and free KL610023 payload | From Cycle 1 to Cycle 6 and End of Treatment(EOT), approximately 12 months
  To characterize the PK of SKB264-ADC, SKB264 TAB, and free KL610023 payload, such as half life
Phase II: Levels of TROP2 expression in tumor tissue | Screening and End of Treatment(EOT), approximately 12 months
  To assess levels of TROP2 expression in tumor tissue and correlation of those levels with responses and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon Ahnert, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (109):
- United States (10):
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - University of California Los Angeles, Los Angeles, California
  - Florida Cancer Specialists and Research Institute, Sarasota, Florida
  - START MidWest, Grand Rapids, Michigan
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - MUHC,Glen - Women's Health Research Unit, Montreal, Quebec
- Chile (3):
  - Centro de Estudios Clínicos SAGA, Providencia
  - Centro de Investigacion Clinica Bradford Hill, Santiago
  - Pontificia Universidad Catolica de Chile - CICUC, Santiago
- China (82):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - AnHui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital (301 Hospital), Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hosptital, Chongqing, Chongqing Municipality
  - 900TH Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Uion Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital , Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer prevention Center, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Cancer Center, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang City Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Center Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College Huazhong University Of Science And Technology, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University Of Science And Technology, Wuhan, Hubei
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The first people's hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Obstetrics&Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Neijiang Second People's Hospital, Neijiang, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang University School of Medical Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Gazi University Medical Faculty, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ouyang Q, Rodon J, Liang Y, Wu X, Li Q, Song L, Yan M, Tong Z, Liu Y, Wainberg ZA, Wang Y, Geng C, Ulahannan SV, Yu G, Sharma MR, Wang X, Wang JS, Spira A, Zhao W, Sanborn RE, Cheng Y, Wang X, Liu G, Li Y, Ge J, Chartash E, Akala OO, Yin Y. Results of a phase 1/2 study of sacituzumab tirumotecan in patients with unresectable locally advanced or metastatic solid tumors refractory to standard therapies. J Hematol Oncol. 2025 Jun 6;18(1):61. doi: 10.1186/s13045-025-01705-2. PMID 40481574
- [Derived] Zhao S, Cheng Y, Wang Q, Li X, Liao J, Rodon J, Meng X, Luo Y, Chen Z, Wang W, Yi T, Li Y, Yin Y, Xu H, Yu G, Mi Y, Fan Y, Wainberg ZA, Wang X, Su C, Yu Q, Lai S, Sun L, Zhuang W, Wang X, Yang J, Li Y, Ge J, Li J, Zhang L, Fang W. Sacituzumab tirumotecan in advanced non-small-cell lung cancer with or without EGFR mutations: phase 1/2 and phase 2 trials. Nat Med. 2025 Jun;31(6):1976-1986. doi: 10.1038/s41591-025-03638-2. Epub 2025 Apr 10. PMID 40210967